CLINICAL TRIAL: NCT00112502
Title: A Randomized, Factorial-Design, Phase II Trial of Temozolomide Alone and in Combination With Possible Permutations of Thalidomide, Isotretinoin and/or Celecoxib as Post-Radiation Adjuvant Therapy of Glioblastoma Multiforme
Brief Title: Temozolomide Alone or in Combination With Thalidomide and/or Isotretinoin and/or Celecoxib in Treating Patients Who Have Undergone Radiation Therapy for Glioblastoma Multiforme
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Treatment
Other Study IDs: 2004-0662; MDA-ID-02586; NCI-6636; MDA-2004-0662; CDR0000432954 (Other: NCI); NCI-2009-00076 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2005-06-02; First posted 2005-06-03 (Estimated); Results first posted 2021-10-18 (Actual); Last update posted 2021-10-18 (Actual); Status verified 2021-09

CONDITIONS: Brain and Central Nervous System Tumors; Glioblastoma Multiforme
Keywords: adult giant cell glioblastoma; adult gliosarcoma; adult glioblastoma
MeSH Terms: conditions — Central Nervous System Neoplasms; Glioblastoma; Gliosarcoma | interventions — Celecoxib; Isotretinoin; Temozolomide; Thalidomide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (8):
- Arm I: TMZ (Active Comparator): Oral Temozolomide (TMZ) 150 mg/m^2 once daily on days 1-7 and 15-21.
  Interventions: Drug: Temozolomide
- Arm II: TMZ + Thalidomide (Experimental): Temozolomide as in arm I and oral Thalidomide (Thal) once daily on days 1-28 (starting dose 200 mg).
  Interventions: Drug: Temozolomide; Drug: Thalidomide
- Arm III: TMZ + Isotretinoin (Experimental): Temozolomide as in Arm I and oral Isotretinoin 40 mg/m^2 twice daily on days 1-21.
  Interventions: Drug: Isotretinoin; Drug: Temozolomide
- Arm IV: TMZ + Celecoxib (Experimental): Temozolomide as in arm I and oral Celecoxib 400 mg twice daily on days 1-28.
  Interventions: Drug: Celecoxib; Drug: Temozolomide
- Arm V: TMZ + Thalidomide + Isotretinoin (Experimental): Temozolomide as in arm I, Thalidomide as in arm II, and Isotretinoin as in arm III.
  Interventions: Drug: Isotretinoin; Drug: Temozolomide; Drug: Thalidomide
- Arm VI: TMZ + Thalidomide + Celecoxib (Experimental): Temozolomide as in Arm I, Thalidomide as in Arm II, and Celecoxib as in Arm IV.
  Interventions: Drug: Celecoxib; Drug: Temozolomide; Drug: Thalidomide
- Arm VII: TMZ + Isotretinoin + Celecoxib (Experimental): Temozolomide as in Arm I, Isotretinoin as in Arm III, and Celecoxib as in Arm IV.
  Interventions: Drug: Celecoxib; Drug: Isotretinoin; Drug: Temozolomide
- Arm VIII: TMZ + Thalidomide + Isotretinoin + Celecoxib (Experimental): Temozolomide as in Arm I, Thalidomide as in Arm II, Isotretinoin as in Arm III, and Celecoxib as in Arm IV.
  Interventions: Drug: Celecoxib; Drug: Isotretinoin; Drug: Temozolomide; Drug: Thalidomide

INTERVENTIONS:
Drug: Celecoxib — 400 mg orally twice a day continuous dosing
  Other Names: Celebrex
  Arms: Arm IV: TMZ + Celecoxib; Arm VI: TMZ + Thalidomide + Celecoxib; Arm VII: TMZ + Isotretinoin + Celecoxib; Arm VIII: TMZ + Thalidomide + Isotretinoin + Celecoxib
Drug: Isotretinoin — 40 mg/m^2 orally twice a day (total daily dose = 80 mg/m^2) days 1-21 of a 28 day cycle.
  Other Names: Accutane; 13-Cis-Retinoic Acid
  Arms: Arm III: TMZ + Isotretinoin; Arm V: TMZ + Thalidomide + Isotretinoin; Arm VII: TMZ + Isotretinoin + Celecoxib; Arm VIII: TMZ + Thalidomide + Isotretinoin + Celecoxib
Drug: Temozolomide — 150 mg/m2 orally daily, 7 days on treatment, 7 days off.
  Other Names: Temodar
Drug: Thalidomide — 400 mg orally every day continuous dosing (starting at 200 mg each day and escalating weekly by 100 mg until the maximum dose of 400 mg/day is achieved)
  Other Names: Thalomid
  Arms: Arm II: TMZ + Thalidomide; Arm V: TMZ + Thalidomide + Isotretinoin; Arm VI: TMZ + Thalidomide + Celecoxib; Arm VIII: TMZ + Thalidomide + Isotretinoin + Celecoxib

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as temozolomide, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Thalidomide may stop the growth of glioblastoma multiforme by blocking blood flow to the tumor. Isotretinoin may help cells that are involved in the body's immune response to work better. Celecoxib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. It is not yet known which temozolomide-containing regimen is more effective in treating glioblastoma multiforme.

PURPOSE: This randomized phase II trial is studying eight different temozolomide-containing regimens to compare how well they work in treating patients who have undergone radiation therapy for glioblastoma multiforme.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare the efficacy of adjuvant temozolomide (TMZ) alone or in combination with thalidomide and/or isotretinoin and/or celecoxib, in terms of 6-month progression-free survival, in patients who have undergone radiotherapy for supratentorial glioblastoma multiforme.
* Compare the toxicity of these regimens in these patients.

OUTLINE: This is a randomized, multicenter study. Patients are randomized to 1 of 8 treatment arms.

* Arm I: Patients receive oral temozolomide once daily on days 1-7 and 15-21.
* Arm II: Patients receive temozolomide as in arm I and oral thalidomide once daily on days 1-28.
* Arm III: Patients receive temozolomide as in arm I and oral isotretinoin twice daily on days 1-21.
* Arm IV: Patients receive temozolomide as in arm I and oral celecoxib twice daily on days 1-28.
* Arm V: Patients receive temozolomide as in arm I, thalidomide as in arm II, and isotretinoin as in arm III.
* Arm VI: Patients receive temozolomide as in arm I, thalidomide as in arm II, and celecoxib as in arm IV.
* Arm VII: Patients receive temozolomide as in arm I, isotretinoin as in arm III, and celecoxib as in arm IV.
* Arm VIII: Patients receive temozolomide as in arm I, thalidomide as in arm II, isotretinoin as in arm III, and celecoxib as in arm IV.

In all arms, treatment repeats every 28 days for up to 12 courses in the absence of disease progression or unacceptable toxicity. Patient may receive additional courses of therapy at the discretion of the treating physician.

After completion of study treatment, patients are followed for at least 30 days and then every 3 months thereafter.

PROJECTED ACCRUAL: A total of 180 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed supratentorial glioblastoma multiforme
* Must have undergone a biopsy OR subtotal or gross total resection of the tumor
* Must have completed post-operative (or post-biopsy) radiotherapy within the past 5 weeks

  * No progressive disease after radiotherapy

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* Karnofsky 60-100%

Life expectancy

* Not specified

Hematopoietic

* Absolute neutrophil count ≥ 1,500/mm^3
* Platelet count ≥ 100,000/mm^3

Hepatic

* Serum glutamate pyruvate transaminase (SGPT) < 2 times upper limit of normal (ULN)
* Alkaline phosphatase < 2 times ULN
* Bilirubin ≤ 1.5 mg/dL

Renal

* blood urea nitrogen (BUN) ≤ 1.5 times ULN
* Creatinine ≤ 1.5 times ULN

Immunologic

* No history of allergic reactions attributed to compounds of similar chemical or biological composition to celecoxib or to sulfonamides
* No asthma, urticaria, or allergic reactions to aspirin or other NSAIDs
* No active infection

Gastrointestinal

* No inflammatory bowel disease
* No history of peptic ulcer disease
* No gastrointestinal bleeding within past 3 months

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective double-method contraception during and for 2 months after study participation

  * Fertile female patients randomized to receive thalidomide must use effective double-method contraception for ≥ 4 weeks before, during, and ≥ 4 weeks after completion of study therapy
  * Fertile male patients randomized to receive thalidomide must use effective contraception during and for ≥ 4 weeks after completion of study therapy
* No blood donation (for patients randomized to receive thalidomide)
* No history of any other cancer except nonmelanoma skin cancer or carcinoma in situ of the cervix or cancer that is in complete remission and patient completed all therapy for that disease ≥ 3 years ago
* No other disease that would obscure toxicity or dangerously alter drug metabolism (e.g., severe connective tissue disease)
* No other serious medical illness

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* Prior temozolomide in combination with radiotherapy allowed
* No other prior or concurrent chemotherapy

Endocrine therapy

* Not specified

Radiotherapy

* See Disease Characteristics
* See Chemotherapy

Surgery

* See Disease Characteristics
* No concurrent surgery

Other

* No other concurrent non-steroidal anti-inflammatory drugs (NSAIDs) (for patients randomized to receive celecoxib)
* No other concurrent investigational drugs
* No other concurrent anticancer therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 178 (Actual)
Dates: Start 2005-09; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marta Penas-Prado, MD, Study Chair — M.D. Anderson Cancer Center
Locations (12):
- United States (12):
  - Hembree Mercy Cancer Center at St. Edward Mercy Medical Center, Fort Smith, Arkansas
  - University of Texas MD Anderson Cancer Center at Orlando, Orlando, Florida
  - CCOP - Atlanta Regional, Atlanta, Georgia
  - CCOP - Central Illinois, Decatur, Illinois
  - CCOP - Wichita, Wichita, Kansas
  - CCOP - Grand Rapids, Grand Rapids, Michigan
  - CCOP - Kalamazoo, Kalamazoo, Michigan
  - CCOP - Kansas City, Kansas City, Missouri
  - Cancer Research for the Ozarks, Springfield, Missouri
  - Arthur G. James Cancer Hospital and Richard J. Solove Research Institute at Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - CCOP - Upstate Carolina, Spartanburg, South Carolina
  - University of Texas MD Anderson Cancer Center, Houston, Texas

REFERENCES:
- [Result] Gilbert MR, Gonzalez J, Hunter K, Hess K, Giglio P, Chang E, Puduvalli V, Groves MD, Colman H, Conrad C, Levin V, Woo S, Mahajan A, de Groot J, Yung WK. A phase I factorial design study of dose-dense temozolomide alone and in combination with thalidomide, isotretinoin, and/or celecoxib as postchemoradiation adjuvant therapy for newly diagnosed glioblastoma. Neuro Oncol. 2010 Nov;12(11):1167-72. doi: 10.1093/neuonc/noq100. Epub 2010 Aug 20. PMID 20729242
- [Derived] Penas-Prado M, Hess KR, Fisch MJ, Lagrone LW, Groves MD, Levin VA, De Groot JF, Puduvalli VK, Colman H, Volas-Redd G, Giglio P, Conrad CA, Salacz ME, Floyd JD, Loghin ME, Hsu SH, Gonzalez J, Chang EL, Woo SY, Mahajan A, Aldape KD, Yung WK, Gilbert MR; MD Anderson Community Clinical Oncology Program; Brain Tumor Trials Collaborative. Randomized phase II adjuvant factorial study of dose-dense temozolomide alone and in combination with isotretinoin, celecoxib, and/or thalidomide for glioblastoma. Neuro Oncol. 2015 Feb;17(2):266-73. doi: 10.1093/neuonc/nou155. Epub 2014 Sep 19. PMID 25239666
- See also: University of Texas (UT) MD Anderson Cancer Center Official Website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment Period: September 2005 to February 2011 from various hospitals and institutions representing the Community Clinical Oncology Program (CCOP). A total of 146 participants were accrued at MD Anderson Cancer Center and 32 at the remaining participating sites.
Groups:
- Arm I: TMZ: Oral Temozolomide (TMZ): 150 mg/m^2 once daily on days 1-7 and 15-21.
- Arm II: TMZ + Thalidomide: Oral Temozolomide (TMZ): 150 mg/m^2 once daily on days 1-7 and 15-21.
  Thalidomide: 400 mg orally every day continuous dosing (starting at 200 mg each day and escalating weekly by 100 mg until the maximum dose of 400 mg/day is achieved).
- Arm III: TMZ + Celecoxib: Oral Temozolomide (TMZ): 150 mg/m^2 once daily on days 1-7 and 15-21.
  Celecoxib: 400 mg orally twice a day continuous dosing.
- Arm IV: TMZ + Isotretinoin: Oral Temozolomide (TMZ): 150 mg/m^2 once daily on days 1-7 and 15-21.
  Isotretinoin: 40 mg/m^2 orally twice a day (total daily dose = 80 mg/m^2) days 1-21 of a 28 day cycle.
- Arm V: TMZ + Isotretinoin + Celecoxib: Oral Temozolomide (TMZ): 150 mg/m^2 once daily on days 1-7 and 15-21.
  Celecoxib: 400 mg orally twice a day continuous dosing.
  Isotretinoin: 40 mg/m^2 orally twice a day (total daily dose = 80 mg/m^2) days 1-21 of a 28 day cycle.
- Arm VI: TMZ + Thalidomide + Celecoxib: Oral Temozolomide (TMZ): 150 mg/m^2 once daily on days 1-7 and 15-21.
  Celecoxib: 400 mg orally twice a day continuous dosing.
  Thalidomide: 400 mg orally every day continuous dosing (starting at 200 mg each day and escalating weekly by 100 mg until the maximum dose of 400 mg/day is achieved).
- Arm VII: TMZ + Thalidomide + Isotretinoin: Oral Temozolomide (TMZ): 150 mg/m^2 once daily on days 1-7 and 15-21.
  Isotretinoin: 40 mg/m^2 orally twice a day (total daily dose = 80 mg/m^2) days 1-21 of a 28 day cycle.
  Thalidomide: 400 mg orally every day continuous dosing (starting at 200 mg each day and escalating weekly by 100 mg until the maximum dose of 400 mg/day is achieved).
- Arm VIII: TMZ + Thalidomide + Isotretinoin + Celecoxib: Oral Temozolomide (TMZ): 150 mg/m^2 once daily on days 1-7 and 15-21.
  Celecoxib: 400 mg orally twice a day continuous dosing.
  Isotretinoin: 40 mg/m^2 orally twice a day (total daily dose = 80 mg/m^2) days 1-21 of a 28 day cycle.
  Thalidomide: 400 mg orally every day continuous dosing (starting at 200 mg each day and escalating weekly by 100 mg until the maximum dose of 400 mg/day is achieved).
Period: Overall Study
Arm/Group | Arm I: TMZ | Arm II: TMZ + Thalidomide | Arm III: TMZ + Celecoxib | Arm IV: TMZ + Isotretinoin | Arm V: TMZ + Isotretinoin + Celecoxib | Arm VI: TMZ + Thalidomide + Celecoxib | Arm VII: TMZ + Thalidomide + Isotretinoin | Arm VIII: TMZ + Thalidomide + Isotretinoin + Celecoxib
Started | 22 | 22 | 22 | 22 | 23 | 22 | 23 | 22
Completed | 22 | 21 | 21 | 18 | 21 | 17 | 20 | 15
Not Completed | 0 | 1 | 1 | 4 | 2 | 5 | 3 | 7
Not completed — Withdrawal by Subject | 0 | 1 | 1 | 4 | 2 | 5 | 3 | 7

BASELINE CHARACTERISTICS:
Population: A 178 participants in total were randomized, out of which 23 participants were randomized but not treated because of consent withdrawal with some further difficulties obtaining insurance coverage.
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm I: TMZ | Arm II: TMZ + Thalidomide | Arm III: TMZ + Celecoxib | Arm IV: TMZ + Isotretinoin | Arm V: TMZ + Isotretinoin + Celecoxib | Arm VI: TMZ + Thalidomide + Celecoxib | Arm VII: TMZ + Thalidomide + Isotretinoin | Arm VIII: TMZ + Thalidomide + Isotretinoin + Celecoxib | Total
Number analyzed (Participants) | 22 | 22 | 22 | 22 | 23 | 22 | 23 | 22 | 178
Age, Customized [Number; unit: participants]
  <=19 years: | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
  Between 20 and 59 years: | 17 | 12 | 17 | 14 | 20 | 18 | 15 | 17 | 130
  >=60 years: | 5 | 10 | 5 | 7 | 3 | 4 | 8 | 5 | 47
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 10 | 5 | 8 | 4 | 6 | 6 | 9 | 55
  Male | 15 | 12 | 17 | 14 | 19 | 16 | 17 | 13 | 123
Region of Enrollment [Number; unit: participants]
  United States | 22 | 22 | 22 | 22 | 23 | 22 | 23 | 22 | 178

OUTCOME MEASURES:

1. Primary Outcome: Median Progression-Free Survival (PFS) Comparison of Thalidomide Arms Versus no Thalidomide Arms
Description: Thalidomide versus not Thalidomide analysis: Comparison of median PFS outcome of participants in arms II, VI, VII and VIII, versus participants in arms I, III, IV and V. Median PFS was estimated using the Kaplan-Meier method from time of randomization to time of progression, death, or last follow-up. Progression defined as 25% increase in the sum of products of all measurable lesions over smallest sum observed (over baseline if no decrease) using the same techniques as baseline, OR clear worsening of any evaluable disease, OR appearance of any new lesion/site, OR failure to return for evaluation due to death or deteriorating condition (unless clearly unrelated to this cancer).
Time Frame: Every 2 cycles (1 cycle = 28 days) from randomization until progression of disease, death or last follow-up, up to one year (12 study cycles).
Measure: Median (95% Confidence Interval); unit: months
Groups:
- Thalidomide: Arm II, Arm VI, Arm VII and Arm VIII: Arm II: TMZ + Thalidomide, Arm VI: TMZ + Thalidomide + Celecoxib, Arm VII: TMZ + Thalidomide + Isotretinoin and Arm VIII: TMZ + Thalidomide + Isotretinoin + Celecoxib
  Thalidomide: 400 mg orally every day continuous dosing (starting at 200 mg each day and escalating weekly by 100 mg until the maximum dose of 400 mg/day is achieved).
  Oral Temozolomide (TMZ): 150 mg/m^2 once daily on days 1-7 and 15-21.
  Celecoxib: 400 mg orally twice a day continuous dosing.
  Isotretinoin: 40 mg/m^2 orally twice a day (total daily dose = 80 mg/m^2) days 1-21 of a 28 day cycle.
- No Thalidomide: Arm I, Arm III, Arm IV and Arm V: Arm I: TMZ, Arm III: TMZ + Celecoxib, Arm IV: TMZ + Isotretinoin and Arm V: TMZ + Isotretinoin + Celecoxib
  Oral Temozolomide (TMZ): 150 mg/m^2 once daily on days 1-7 and 15-21.
  Celecoxib: 400 mg orally twice a day continuous dosing.
  Isotretinoin: 40 mg/m^2 orally twice a day (total daily dose = 80 mg/m^2) days 1-21 of a 28 day cycle.
Arm/Group | Thalidomide: Arm II, Arm VI, Arm VII and Arm VIII | No Thalidomide: Arm I, Arm III, Arm IV and Arm V
Number analyzed (Participants) | 70 | 85
months | 7.6 [NA to NA] — 95% Confidence Interval values are not available to be reported as the PI has left the institution and no study team member is present. Sincere efforts were made to obtain the data for reporting, but were unsuccessful | 8.7 [NA to NA] — 95% Confidence Interval values are not available to be reported as the PI has left the institution and no study team member is present. Sincere efforts were made to obtain the data for reporting, but were unsuccessful
Statistical Analysis 1: Comparison: Thalidomide: Arm II, Arm VI, Arm VII and Arm VIII vs No Thalidomide: Arm I, Arm III, Arm IV and Arm V; Test type: Superiority or Other; Hazard Ratio (HR) = 1.2, 95% CI 2-sided [0.8 to 1.7]

2. Primary Outcome: Median Progression-Free Survival (PFS) Comparison of Celecoxib Arms Versus no Celecoxib Arms
Description: Celecoxib versus not Celecoxib analysis: We compared the median PFS outcome of participants in arms III, V, VI and VIII, versus participants in arms I, II, IV and VII. Median PFS was estimated using the Kaplan-Meier method from time of randomization to time of progression, death, or last follow-up. Progression defined as 25% increase in the sum of products of all measurable lesions over smallest sum observed (over baseline if no decrease) using the same techniques as baseline, OR clear worsening of any evaluable disease, OR appearance of any new lesion/site, OR failure to return for evaluation due to death or deteriorating condition (unless clearly unrelated to this cancer).
Time Frame: Every 2 cycles (1 cycle = 28 days) from randomization until progression of disease, death or last follow-up.
Measure: Median (95% Confidence Interval); unit: months
Groups:
- Celecoxib: Arm III, Arm V, Arm VI and Arm VIII: Arm III: TMZ + Celecoxib, Arm V: TMZ + Isotretinoin + Celecoxib, Arm VI: TMZ + Thalidomide + Celecoxib and Arm VIII: TMZ + Thalidomide + Isotretinoin + Celecoxib
  Thalidomide: 400 mg orally every day continuous dosing (starting at 200 mg each day and escalating weekly by 100 mg until the maximum dose of 400 mg/day is achieved).
  Oral Temozolomide (TMZ): 150 mg/m^2 once daily on days 1-7 and 15-21.
  Celecoxib: 400 mg orally twice a day continuous dosing.
  Isotretinoin: 40 mg/m^2 orally twice a day (total daily dose = 80 mg/m^2) days 1-21 of a 28 day cycle.
- No Celecoxib: Arm I, Arm II, Arm IV and Arm VII: Arm I: TMZ, Arm II: TMZ + Thalidomide, Arm IV: TMZ + Isotretinoin and Arm VII: TMZ + Thalidomide + Isotretinoin.
  Thalidomide: 400 mg orally every day continuous dosing (starting at 200 mg each day and escalating weekly by 100 mg until the maximum dose of 400 mg/day is achieved).
  Oral Temozolomide (TMZ): 150 mg/m^2 once daily on days 1-7 and 15-21.
  Isotretinoin: 40 mg/m^2 orally twice a day (total daily dose = 80 mg/m^2) days 1-21 of a 28 day cycle.
Arm/Group | Celecoxib: Arm III, Arm V, Arm VI and Arm VIII | No Celecoxib: Arm I, Arm II, Arm IV and Arm VII
Number analyzed (Participants) | 74 | 81
months | 8.3 [NA to NA] — 95% Confidence Interval values are not available to be reported as the PI has left the institution and no study team member is present. Sincere efforts were made to obtain the data for reporting, but were unsuccessful | 7.4 [NA to NA] — 95% Confidence Interval values are not available to be reported as the PI has left the institution and no study team member is present. Sincere efforts were made to obtain the data for reporting, but were unsuccessful
Statistical Analysis 1: Comparison: Celecoxib: Arm III, Arm V, Arm VI and Arm VIII vs No Celecoxib: Arm I, Arm II, Arm IV and Arm VII; Test type: Superiority or Other; Hazard Ratio (HR) = 0.8, 95% CI 2-sided [0.6 to 1.2]

3. Primary Outcome: Median Progression-Free Survival (PFS) Comparison of Isotretinoin Arms Versus no Isotretinoin Arms
Description: Isotretinoin versus not Isotretinoin analysis: We compared the median PFS outcome of participants in arms IV, V, VII and VIII, versus participants in arms I, II, III and VI. Median PFS was estimated using the Kaplan-Meier method from time of randomization to time of progression, death, or last follow-up. Progression defined as 25% increase in the sum of products of all measurable lesions over smallest sum observed (over baseline if no decrease) using the same techniques as baseline, OR clear worsening of any evaluable disease, OR appearance of any new lesion/site, OR failure to return for evaluation due to death or deteriorating condition (unless clearly unrelated to this cancer).
Time Frame: Every 2 cycles (1 cycle = 28 days) from randomization until progression of disease, death or last follow-up.
Measure: Median (95% Confidence Interval); unit: months
Groups:
- Isotretinoin: Arm IV, Arm V, Arm VII and Arm VIII: Arm IV: TMZ + Isotretinoin, Arm V: TMZ + Isotretinoin + Celecoxib, Arm VII: TMZ + Thalidomide + Isotretinoin and Arm VIII: TMZ + Thalidomide + Isotretinoin + Celecoxib
  Thalidomide: 400 mg orally every day continuous dosing (starting at 200 mg each day and escalating weekly by 100 mg until the maximum dose of 400 mg/day is achieved).
  Oral Temozolomide (TMZ): 150 mg/m^2 once daily on days 1-7 and 15-21.
  Celecoxib: 400 mg orally twice a day continuous dosing.
  Isotretinoin: 40 mg/m^2 orally twice a day (total daily dose = 80 mg/m^2) days 1-21 of a 28 day cycle.
- No Isotretinoin: Arm I, Arm II, Arm III and Arm VI: Arm I: TMZ, Arm II: TMZ + Thalidomide, Arm III: TMZ + Celecoxib and Arm VI: TMZ + Thalidomide + Celecoxib
  Thalidomide: 400 mg orally every day continuous dosing (starting at 200 mg each day and escalating weekly by 100 mg until the maximum dose of 400 mg/day is achieved).
  Oral Temozolomide (TMZ): 150 mg/m^2 once daily on days 1-7 and 15-21.
  Celecoxib: 400 mg orally twice a day continuous dosing.
Arm/Group | Isotretinoin: Arm IV, Arm V, Arm VII and Arm VIII | No Isotretinoin: Arm I, Arm II, Arm III and Arm VI
Number analyzed (Participants) | 74 | 81
months | 6.6 [NA to NA] — 95% Confidence Interval values are not available to be reported as the PI has left the institution and no study team member is present. Sincere efforts were made to obtain the data for reporting, but were unsuccessful | 9.1 [NA to NA] — 95% Confidence Interval values are not available to be reported as the PI has left the institution and no study team member is present. Sincere efforts were made to obtain the data for reporting, but were unsuccessful
Statistical Analysis 1: Comparison: Isotretinoin: Arm IV, Arm V, Arm VII and Arm VIII vs No Isotretinoin: Arm I, Arm II, Arm III and Arm VI; Test type: Superiority or Other; Hazard Ratio (HR) = 1.3, 95% CI 2-sided [0.9 to 1.8]

4. Secondary Outcome: Median Progression-Free Survival (PFS) Comparison of Doublet Versus Triplet Therapy
Description: Doublet (2 agents) versus Triplet (3 agents) therapy analysis: We compared the median PFS outcome of participants in arms II, III, IV, versus participants in arms V, VI and VII. Median PFS was estimated using the Kaplan-Meier method from time of randomization to time of progression, death, or last follow-up. Progression defined as 25% increase in the sum of products of all measurable lesions over smallest sum observed (over baseline if no decrease) using the same techniques as baseline, OR clear worsening of any evaluable disease, OR appearance of any new lesion/site, OR failure to return for evaluation due to death or deteriorating condition (unless clearly unrelated to this cancer).
Time Frame: Every 2 cycles (1 cycle = 28 days) from randomization until progression of disease, death or last follow-up.
Measure: Median (95% Confidence Interval); unit: months
Groups:
- Doublet (2 Agents): Arm II, Arm III and Arm IV: Arm II: TMZ + Thalidomide, Arm III: TMZ + Celecoxib and Arm IV: TMZ + Isotretinoin
  Oral Temozolomide (TMZ): 150 mg/m^2 once daily on days 1-7 and 15-21.
  Thalidomide: 400 mg orally every day continuous dosing (starting at 200 mg each day and escalating weekly by 100 mg until the maximum dose of 400 mg/day is achieved).
  Celecoxib: 400 mg orally twice a day continuous dosing.
  Isotretinoin: 40 mg/m^2 orally twice a day (total daily dose = 80 mg/m^2) days 1-21 of a 28 day cycle.
- Triplet (3 Agents): Arm V, Arm VI and Arm VII: Arm V: TMZ + Isotretinoin + Celecoxib, Arm VI: TMZ + Thalidomide + Celecoxib and Arm VII: Thalidomide + Celecoxib + Isotretinoin
  Oral Temozolomide (TMZ): 150 mg/m^2 once daily on days 1-7 and 15-21.
  Thalidomide: 400 mg orally every day continuous dosing (starting at 200 mg each day and escalating weekly by 100 mg until the maximum dose of 400 mg/day is achieved).
  Celecoxib: 400 mg orally twice a day continuous dosing.
  Isotretinoin: 40 mg/m^2 orally twice a day (total daily dose = 80 mg/m^2) days 1-21 of a 28 day cycle.
Arm/Group | Doublet (2 Agents): Arm II, Arm III and Arm IV | Triplet (3 Agents): Arm V, Arm VI and Arm VII
Number analyzed (Participants) | 60 | 58
months | 8.3 [NA to NA] — 95% Confidence Interval values are not available to be reported as the PI has left the institution and no study team member is present. Sincere efforts were made to obtain the data for reporting, but were unsuccessful | 8.2 [NA to NA] — 95% Confidence Interval values are not available to be reported as the PI has left the institution and no study team member is present. Sincere efforts were made to obtain the data for reporting, but were unsuccessful
Statistical Analysis 1: Comparison: Doublet (2 Agents): Arm II, Arm III and Arm IV vs Triplet (3 Agents): Arm V, Arm VI and Arm VII; Test type: Superiority or Other; Hazard Ratio (HR) = 0.9, 95% CI 2-sided [0.6 to 1.3]

5. Secondary Outcome: Median Progression-Free Survival (PFS) of Individual Arms
Description: Median PFS was estimated using the Kaplan-Meier method from time of randomization to time of progression, death, or last follow-up. Progression defined as 25% increase in the sum of products of all measurable lesions over smallest sum observed (over baseline if no decrease) using the same techniques as baseline, OR clear worsening of any evaluable disease, OR appearance of any new lesion/site, OR failure to return for evaluation due to death or deteriorating condition (unless clearly unrelated to this cancer).
Time Frame: Every 2 cycles (1 cycle = 28 days) from randomization until progression of disease, death or last follow-up.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm I: TMZ | Arm II: TMZ + Thalidomide | Arm III: TMZ + Celecoxib | Arm IV: TMZ + Isotretinoin | Arm V: TMZ + Isotretinoin + Celecoxib | Arm VI: TMZ + Thalidomide + Celecoxib | Arm VII: TMZ + Thalidomide + Isotretinoin | Arm VIII: TMZ + Thalidomide + Isotretinoin + Celecoxib
Number analyzed (Participants) | 22 | 18 | 21 | 21 | 21 | 20 | 17 | 15
months | 10.5 [NA to NA] — 95% Confidence Interval values are not available to be reported as the PI has left the institution and no study team member is present. Sincere efforts were made to obtain the data for reporting, but were unsuccessful | 7.7 [NA to NA] — 95% Confidence Interval values are not available to be reported as the PI has left the institution and no study team member is present. Sincere efforts were made to obtain the data for reporting, but were unsuccessful | 13.4 [NA to NA] — 95% Confidence Interval values are not available to be reported as the PI has left the institution and no study team member is present. Sincere efforts were made to obtain the data for reporting, but were unsuccessful | 6.5 [NA to NA] — 95% Confidence Interval values are not available to be reported as the PI has left the institution and no study team member is present. Sincere efforts were made to obtain the data for reporting, but were unsuccessful | 11.6 [NA to NA] — 95% Confidence Interval values are not available to be reported as the PI has left the institution and no study team member is present. Sincere efforts were made to obtain the data for reporting, but were unsuccessful | 7.9 [NA to NA] — 95% Confidence Interval values are not available to be reported as the PI has left the institution and no study team member is present. Sincere efforts were made to obtain the data for reporting, but were unsuccessful | 6.2 [NA to NA] — 95% Confidence Interval values are not available to be reported as the PI has left the institution and no study team member is present. Sincere efforts were made to obtain the data for reporting, but were unsuccessful | 5.8 [NA to NA] — 95% Confidence Interval values are not available to be reported as the PI has left the institution and no study team member is present. Sincere efforts were made to obtain the data for reporting, but were unsuccessful

6. Secondary Outcome: Median Overall Survival (OS) Comparison of Thalidomide Arms Versus no Thalidomide Arms
Description: Thalidomide versus not Thalidomide analysis: We compared the median OS outcome of participants in arms II, VI, VII and VIII, versus participants in arms I, III, IV and V. Median OS was estimated using the Kaplan-Meier method from time of randomization to time of progression, death, or last follow-up. Progression defined as 25% increase in the sum of products of all measurable lesions over smallest sum observed (over baseline if no decrease) using the same techniques as baseline, OR clear worsening of any evaluable disease, OR appearance of any new lesion/site, OR failure to return for evaluation due to death or deteriorating condition (unless clearly unrelated to this cancer).
Time Frame: Every 3 months from randomization until progression of disease, death or last follow-up.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Thalidomide: Arm II, Arm VI, Arm VII and Arm VIII | No Thalidomide: Arm I, Arm III, Arm IV and Arm V
Number analyzed (Participants) | 70 | 85
months | 18.3 [NA to NA] — 95% Confidence Interval values are not available to be reported as the PI has left the institution and no study team member is present. Sincere efforts were made to obtain the data for reporting, but were unsuccessful | 17.4 [NA to NA] — 95% Confidence Interval values are not available to be reported as the PI has left the institution and no study team member is present. Sincere efforts were made to obtain the data for reporting, but were unsuccessful
Statistical Analysis 1: Comparison: Thalidomide: Arm II, Arm VI, Arm VII and Arm VIII vs No Thalidomide: Arm I, Arm III, Arm IV and Arm V; Test type: Superiority or Other; Hazard Ratio (HR) = 1.0, 95% CI 2-sided [0.7 to 1.5]

7. Secondary Outcome: Median Overall Survival (OS) Comparison of Celecoxib Arms Versus no Celecoxib Arms
Description: Celecoxib versus not Celecoxib analysis: We compared the median OS outcome of participants in arms III, V, VI and VIII, versus participants in arms I, II, IV and VII. Median OS was estimated using the Kaplan-Meier method from time of randomization to time of progression, death, or last follow-up. Progression defined as 25% increase in the sum of products of all measurable lesions over smallest sum observed (over baseline if no decrease) using the same techniques as baseline, OR clear worsening of any evaluable disease, OR appearance of any new lesion/site, OR failure to return for evaluation due to death or deteriorating condition (unless clearly unrelated to this cancer).
Time Frame: Every 3 months from randomization until progression of disease, death or last follow-up.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Celecoxib: Arm III, Arm V, Arm VI and Arm VIII | No Celecoxib: Arm I, Arm II, Arm IV and Arm VII
Number analyzed (Participants) | 74 | 81
months | 20.2 [NA to NA] — 95% Confidence Interval values are not available to be reported as the PI has left the institution and no study team member is present. Sincere efforts were made to obtain the data for reporting, but were unsuccessful | 17.1 [NA to NA] — 95% Confidence Interval values are not available to be reported as the PI has left the institution and no study team member is present. Sincere efforts were made to obtain the data for reporting, but were unsuccessful
Statistical Analysis 1: Comparison: Celecoxib: Arm III, Arm V, Arm VI and Arm VIII vs No Celecoxib: Arm I, Arm II, Arm IV and Arm VII; Test type: Superiority or Other; Hazard Ratio (HR) = 0.8, 95% CI 2-sided [0.5 to 1.2]

8. Secondary Outcome: Median Overall Survival (OS) Comparison of Isotretinoin Arms Versus no Isotretinoin Arms
Description: Isotretinoin versus not Isotretinoin analysis: We compared the median OS outcome of participants in arms IV, V, VII and VIII, versus participants in arms I, II, III and VI. Median OS was estimated using the Kaplan-Meier method from time of randomization to time of progression, death, or last follow-up. Progression defined as 25% increase in the sum of products of all measurable lesions over smallest sum observed (over baseline if no decrease) using the same techniques as baseline, OR clear worsening of any evaluable disease, OR appearance of any new lesion/site, OR failure to return for evaluation due to death or deteriorating condition (unless clearly unrelated to this cancer).
Time Frame: Every 3 months from randomization until progression of disease, death or last follow-up.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Isotretinoin: Arm IV, Arm V, Arm VII and ARM VIII | No Isotretinoin: Arm I, Arm II, Arm III and ARM VI
Number analyzed (Participants) | 74 | 81
months | 17.1 [NA to NA] — 95% Confidence Interval values are not available to be reported as the PI has left the institution and no study team member is present. Sincere efforts were made to obtain the data for reporting, but were unsuccessful | 19.9 [NA to NA] — 95% Confidence Interval values are not available to be reported as the PI has left the institution and no study team member is present. Sincere efforts were made to obtain the data for reporting, but were unsuccessful
Statistical Analysis 1: Comparison: Isotretinoin: Arm IV, Arm V, Arm VII and ARM VIII vs No Isotretinoin: Arm I, Arm II, Arm III and ARM VI; Test type: Superiority or Other; Hazard Ratio (HR) = 1.2, 95% CI 2-sided [0.8 to 1.8]

9. Secondary Outcome: Median Overall Survival (OS) Comparison of Doublet Versus Triplet Therapy
Description: Doublet (2 agents) versus Triplet (3 agents) therapy analysis: We compared the median OS outcome of participants in arms II, III, IV, versus participants in arms V, VI and VII. Median OS was estimated using the Kaplan-Meier method from time of randomization to time of progression, death, or last follow-up. Progression defined as 25% increase in the sum of products of all measurable lesions over smallest sum observed (over baseline if no decrease) using the same techniques as baseline, OR clear worsening of any evaluable disease, OR appearance of any new lesion/site, OR failure to return for evaluation due to death or deteriorating condition (unless clearly unrelated to this cancer).
Time Frame: Every 3 months from randomization until progression of disease, death or last follow-up.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Doublet (2 Agents): Arm II, Arm III and Arm IV | Triplet (3 Agents): Arm V, Arm VI and Arm VII
Number analyzed (Participants) | 60 | 58
months | 17.0 [NA to NA] — 95% Confidence Interval values are not available to be reported as the PI has left the institution and no study team member is present. Sincere efforts were made to obtain the data for reporting, but were unsuccessful | 20.1 [NA to NA] — 95% Confidence Interval values are not available to be reported as the PI has left the institution and no study team member is present. Sincere efforts were made to obtain the data for reporting, but were unsuccessful
Statistical Analysis 1: Comparison: Doublet (2 Agents): Arm II, Arm III and Arm IV vs Triplet (3 Agents): Arm V, Arm VI and Arm VII; Test type: Superiority or Other; Hazard Ratio (HR) = 0.7, 95% CI 2-sided [0.5 to 1.1]

10. Secondary Outcome: Overall Survival of Individual Arms
Description: Overall Survival (OS) was estimated using the Kaplan-Meier method from time of randomization to time of progression, death, or last follow-up. Progression defined as 25% increase in the sum of products of all measurable lesions over smallest sum observed (over baseline if no decrease) using the same techniques as baseline, OR clear worsening of any evaluable disease, OR appearance of any new lesion/site, OR failure to return for evaluation due to death or deteriorating condition (unless clearly unrelated to this cancer).
Time Frame: Every 3 months from randomization until progression of disease, death or last follow-up.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm I: TMZ | Arm II: TMZ + Thalidomide | Arm III: TMZ + Celecoxib | Arm IV: TMZ + Isotretinoin | Arm V: TMZ + Isotretinoin + Celecoxib | Arm VI: TMZ + Thalidomide + Celecoxib | Arm VII: TMZ + Thalidomide + Isotretinoin | Arm VIII: TMZ + Thalidomide + Isotretinoin + Celecoxib
Number analyzed (Participants) | 22 | 18 | 21 | 21 | 21 | 20 | 17 | 15
months | 21.2 [NA to NA] — 95% Confidence Interval values are not available to be reported as the PI has left the institution and no study team member is present. Sincere efforts were made to obtain the data for reporting, but were unsuccessful | 17.4 [NA to NA] — 95% Confidence Interval values are not available to be reported as the PI has left the institution and no study team member is present. Sincere efforts were made to obtain the data for reporting, but were unsuccessful | 18.1 [NA to NA] — 95% Confidence Interval values are not available to be reported as the PI has left the institution and no study team member is present. Sincere efforts were made to obtain the data for reporting, but were unsuccessful | 11.7 [NA to NA] — 95% Confidence Interval values are not available to be reported as the PI has left the institution and no study team member is present. Sincere efforts were made to obtain the data for reporting, but were unsuccessful | 23.1 [NA to NA] — 95% Confidence Interval values are not available to be reported as the PI has left the institution and no study team member is present. Sincere efforts were made to obtain the data for reporting, but were unsuccessful | 20.2 [NA to NA] — 95% Confidence Interval values are not available to be reported as the PI has left the institution and no study team member is present. Sincere efforts were made to obtain the data for reporting, but were unsuccessful | 17.9 [NA to NA] — 95% Confidence Interval values are not available to be reported as the PI has left the institution and no study team member is present. Sincere efforts were made to obtain the data for reporting, but were unsuccessful | 18.5 [NA to NA] — 95% Confidence Interval values are not available to be reported as the PI has left the institution and no study team member is present. Sincere efforts were made to obtain the data for reporting, but were unsuccessful

ADVERSE EVENTS:
Time Frame: Adverse Events (AEs) and Serious Adverse Events (SAEs) were collected from study drug administration to time of progression, death, or last follow-up,1 year", "Adverse Events (AEs) and Serious Adverse Events (SAEs) were collected from study drug administration to time of progression, death, or last follow-up, up to 5 years.
Arm/Group | Arm I: TMZ | Arm II: TMZ + Thalidomide | Arm III: TMZ + Celecoxib | Arm IV: TMZ + Isotretinoin | Arm V: TMZ + Isotretinoin + Celecoxib | Arm VI: TMZ + Thalidomide + Celecoxib | Arm VII: TMZ + Thalidomide + Isotretinoin | Arm VIII: TMZ + Thalidomide + Isotretinoin + Celecoxib
Serious Adverse Events (participants affected / at risk) | 11/22 | 9/21 | 7/21 | 8/18 | 12/21 | 15/17 | 8/20 | 7/15
Other Adverse Events (participants affected / at risk) | 22/22 | 21/21 | 21/21 | 18/18 | 21/21 | 17/17 | 20/20 | 15/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I: TMZ (N=22) | Arm II: TMZ + Thalidomide (N=21) | Arm III: TMZ + Celecoxib (N=21) | Arm IV: TMZ + Isotretinoin (N=18) | Arm V: TMZ + Isotretinoin + Celecoxib (N=21) | Arm VI: TMZ + Thalidomide + Celecoxib (N=17) | Arm VII: TMZ + Thalidomide + Isotretinoin (N=20) | Arm VIII: TMZ + Thalidomide + Isotretinoin + Celecoxib (N=15)
Lymphopenia (Blood and lymphatic system disorders) | 10 (10) | 5 (5) | 5 (5) | 5 (5) | 11 (11) | 10 (10) | 3 (3) | 4 (4)
Platelets (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Thrombosis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 1 (1)
Leukocytes (Blood and lymphatic system disorders) | 0 (0) | 2 (2) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Neutrophils (Blood and lymphatic system disorders) | 0 (0) | 3 (3) | 0 (0) | 2 (2) | 0 (0) | 2 (2) | 3 (3) | 1 (1)
Pyramidal Tract Dysfunction (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gait/Walking (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Death (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Fatigue (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hemoglobin (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperkalemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperglycemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Obesity (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sinus Bradycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pulmonary Embolism (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Erythema Multiforme (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I: TMZ (N=22) | Arm II: TMZ + Thalidomide (N=21) | Arm III: TMZ + Celecoxib (N=21) | Arm IV: TMZ + Isotretinoin (N=18) | Arm V: TMZ + Isotretinoin + Celecoxib (N=21) | Arm VI: TMZ + Thalidomide + Celecoxib (N=17) | Arm VII: TMZ + Thalidomide + Isotretinoin (N=20) | Arm VIII: TMZ + Thalidomide + Isotretinoin + Celecoxib (N=15)
Leukocytes (Blood and lymphatic system disorders) | 16 (54) | 14 (28) | 16 (43) | 15 (34) | 16 (66) | 17 (35) | 11 (36) | 14 (32)
Lymphopenia (Blood and lymphatic system disorders) | 22 (99) | 21 (35) | 21 (70) | 18 (50) | 21 (74) | 17 (69) | 12 (23) | 12 (17)
Neutrophils (Blood and lymphatic system disorders) | 13 (37) | 11 (25) | 9 (30) | 10 (21) | 11 (19) | 17 (24) | 7 (27) | 12 (22)
Platelets (Blood and lymphatic system disorders) | 13 (35) | 5 (8) | 12 (28) | 13 (17) | 11 (31) | 14 (26) | 9 (22) | 11 (14)
Fatigue (General disorders) | 19 (27) | 13 (16) | 16 (20) | 14 (15) | 17 (20) | 17 (26) | 14 (16) | 14 (16)
Rash (Skin and subcutaneous tissue disorders) | 8 (8) | 5 (5) | 6 (10) | 1 (1) | 4 (4) | 11 (12) | 6 (7) | 4 (4)
Anorexia (Gastrointestinal disorders) | 8 (9) | 2 (2) | 3 (3) | 7 (10) | 3 (3) | 9 (10) | 4 (4) | 3 (3)
Infection (Infections and infestations) | 1 (1) | 3 (3) | 0 (0) | 1 (1) | 3 (3) | 2 (2) | 1 (1) | 1 (1) — Normal ANC or Grade 1 or 2 neutrophils
Muscle Weakness (Musculoskeletal and connective tissue disorders) | 11 (16) | 5 (5) | 9 (10) | 11 (14) | 7 (7) | 11 (14) | 4 (4) | 4 (5)
Syncope (Nervous system disorders) | 1 (1) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Hemoglobin (Blood and lymphatic system disorders) | 16 (39) | 8 (12) | 17 (39) | 14 (31) | 15 (39) | 17 (45) | 9 (25) | 11 (26)
Hyperglycemia (Metabolism and nutrition disorders) | 18 (35) | 8 (10) | 17 (38) | 10 (20) | 11 (17) | 9 (18) | 10 (20) | 9 (10)
Depression (Psychiatric disorders) | 3 (4) | 2 (2) | 2 (2) | 4 (5) | 8 (8) | 5 (6) | 2 (2) | 4 (4)
Pruritus (Skin and subcutaneous tissue disorders) | 4 (4) | 0 (0) | 3 (3) | 3 (3) | 2 (2) | 1 (2) | 2 (2) | 2 (2)
Amylase (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1) | 2 (4) | 5 (15) | 0 (0) | 1 (2) | 0 (0)
Hypertriglyceridemia (Metabolism and nutrition disorders) | 6 (7) | 7 (7) | 7 (7) | 10 (21) | 16 (30) | 3 (3) | 11 (17) | 11 (14)
Hypoalbuminemia (Metabolism and nutrition disorders) | 2 (3) | 3 (8) | 3 (4) | 3 (3) | 2 (3) | 4 (5) | 2 (2) | 4 (5)
Hypophosphatemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 5 (5) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Lipase (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1) | 7 (8) | 9 (23) | 1 (1) | 3 (3) | 3 (5)
Pain (General disorders) | 1 (1) | 2 (2) | 2 (2) | 5 (7) | 1 (1) | 4 (4) | 4 (5) | 5 (6) — Extremity-limb
Speech Impairment (General disorders) | 2 (2) | 6 (6) | 4 (4) | 4 (4) | 7 (7) | 4 (5) | 8 (8) | 1 (1)
Opportunistic Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1) | 1 (1) | 4 (5) | 3 (4) | 5 (6) | 3 (5) | 2 (2)
Hypokalemia (Metabolism and nutrition disorders) | 3 (4) | 1 (1) | 3 (4) | 3 (3) | 4 (6) | 4 (5) | 4 (7) | 3 (4)
ALT, SGPT (Hepatobiliary disorders) | 6 (7) | 5 (6) | 8 (14) | 7 (7) | 6 (9) | 4 (5) | 8 (8) | 7 (9)
AST, SGOT (Hepatobiliary disorders) | 4 (4) | 5 (8) | 9 (10) | 3 (3) | 5 (5) | 6 (10) | 6 (6) | 6 (7)
Sinus Bradycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Thrombosis (Vascular disorders) | 4 (5) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 1 (1) | 0 (0)
Weight Loss (General disorders) | 10 (11) | 1 (1) | 5 (5) | 3 (4) | 7 (8) | 4 (4) | 4 (4) | 5 (5)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 4 (4) | 0 (0)
Fever (General disorders) | 4 (5) | 1 (1) | 0 (0) | 3 (5) | 1 (1) | 2 (2) | 3 (4) | 2 (2) — Absence of Neutropenia
Headache (Nervous system disorders) | 10 (13) | 9 (11) | 9 (9) | 14 (15) | 12 (17) | 8 (10) | 13 (16) | 8 (9)
Constipation (Gastrointestinal disorders) | 13 (13) | 11 (11) | 9 (9) | 11 (12) | 8 (8) | 12 (14) | 10 (10) | 8 (8)
Hypercholesteremia (Metabolism and nutrition disorders) | 9 (12) | 6 (6) | 3 (3) | 13 (17) | 16 (22) | 4 (4) | 8 (8) | 9 (10)
Dizziness (Nervous system disorders) | 7 (7) | 6 (6) | 9 (10) | 6 (6) | 8 (9) | 11 (13) | 9 (9) | 3 (3)
Dry Skin (Skin and subcutaneous tissue disorders) | 3 (3) | 2 (2) | 4 (4) | 11 (13) | 19 (19) | 9 (9) | 9 (9) | 10 (10)
Ataxia (Nervous system disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 4 (4) | 5 (5) | 2 (2) | 1 (1)
Pyramidal Tract Dysfunction (Nervous system disorders) | 10 (10) | 5 (5) | 7 (7) | 6 (6) | 7 (7) | 8 (8) | 8 (8) | 4 (4)
Alkaline Phosphatase (Metabolism and nutrition disorders) | 6 (14) | 2 (2) | 2 (4) | 4 (5) | 5 (11) | 2 (2) | 2 (2) | 1 (1)
Allergic Reaction (Immune system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Allergic Rhinitis (Immune system disorders) | 2 (2) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 3 (3) | 4 (4) | 5 (5) | 4 (4) | 5 (5) | 1 (1) | 3 (3) | 6 (6)
Rhinitis (Immune system disorders) | 2 (3) | 0 (0) | 1 (1) | 1 (1) | 3 (3) | 2 (4) | 4 (4) | 2 (2)
Hearing Loss (Ear and labyrinth disorders) | 1 (1) | 1 (1) | 5 (5) | 3 (3) | 1 (1) | 3 (3) | 3 (3) | 2 (2)
Left Ear Drainage (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Low Bicarbonate (Metabolism and nutrition disorders) | 2 (2) | 2 (5) | 2 (2) | 7 (7) | 2 (2) | 1 (1) | 1 (1) | 2 (2)
Hyperbilirubinemia (Metabolism and nutrition disorders) | 2 (3) | 3 (3) | 3 (5) | 3 (7) | 3 (6) | 1 (1) | 1 (1) | 3 (3)
Anemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 2 (3) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 2 (4)
Hematocrit (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blurred Vision (Eye disorders) | 4 (6) | 1 (1) | 4 (4) | 2 (2) | 4 (4) | 4 (4) | 3 (4) | 4 (4)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bruising (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Supraventricular Arrhythmia-Sinus Tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
CO2 Serum High (Blood and lymphatic system disorders) | 4 (5) | 2 (2) | 5 (6) | 1 (1) | 2 (2) | 4 (7) | 4 (4) | 2 (2)
Cognitive Disturbance (Nervous system disorders) | 6 (7) | 4 (4) | 7 (7) | 5 (5) | 5 (5) | 5 (5) | 5 (5) | 3 (3)
Colitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Confusion (Nervous system disorders) | 3 (4) | 0 (0) | 4 (5) | 5 (5) | 1 (1) | 4 (4) | 4 (4) | 3 (3)
Cough (Respiratory, thoracic and mediastinal disorders) | 8 (10) | 3 (3) | 3 (4) | 7 (8) | 3 (4) | 2 (2) | 6 (8) | 3 (4)
Creatinine (Metabolism and nutrition disorders) | 6 (7) | 3 (3) | 2 (2) | 5 (5) | 4 (6) | 5 (5) | 4 (4) | 2 (3)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 3 (5) | 4 (4) | 1 (1) | 4 (4) | 5 (6) | 3 (3)
Xerostomia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 2 (2) | 1 (1) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Edema (Blood and lymphatic system disorders) | 4 (4) | 2 (2) | 6 (6) | 2 (2) | 3 (4) | 6 (9) | 3 (4) | 6 (6) — Limb
Erectile Dysfunction (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gait/Walking (Musculoskeletal and connective tissue disorders) | 5 (5) | 5 (5) | 7 (8) | 6 (7) | 6 (7) | 8 (8) | 10 (10) | 4 (4)
Bloating (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Hypoglycemia (Metabolism and nutrition disorders) | 3 (3) | 0 (0) | 5 (5) | 1 (2) | 1 (1) | 1 (1) | 2 (2) | 0 (0)
Heartburn (Gastrointestinal disorders) | 1 (1) | 1 (1) | 2 (2) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 2 (2)
Hot Flashes (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hemorrhage (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 3 (4) | 1 (2) | 0 (0) | 3 (3) | 1 (1)
Hypercalcemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Hyperkalemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 3 (3) | 1 (1) | 4 (6) | 1 (1) | 2 (2) | 2 (3)
Hypermagnesemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Cardiac disorders) | 4 (6) | 4 (4) | 1 (2) | 4 (4) | 2 (2) | 1 (1) | 4 (5) | 2 (2)
Hyperuricemia (Metabolism and nutrition disorders) | 5 (5) | 1 (1) | 5 (6) | 2 (2) | 6 (9) | 1 (1) | 1 (2) | 0 (0)
Hypocalcemia (Metabolism and nutrition disorders) | 1 (1) | 1 (3) | 3 (7) | 1 (1) | 2 (2) | 3 (3) | 2 (2) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 5 (6) | 3 (4) | 2 (2) | 3 (3) | 4 (6) | 1 (1) | 0 (0) | 1 (1)
Hypotension (Cardiac disorders) | 1 (1) | 1 (1) | 2 (2) | 2 (2) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Upper Respiratory Infection (Respiratory, thoracic and mediastinal disorders) | 3 (6) | 3 (3) | 0 (0) | 3 (3) | 1 (1) | 1 (1) | 1 (1) | 2 (2)
Cellulitis (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Herpes (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infection with Unknown ANC (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Vagina - yeast
Gingivitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Urinary Tract Infection (Renal and urinary disorders) | 1 (1) | 1 (1) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Shingles (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Infection with Normal ANC (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — Eye
Infection with Normal ANC (Infections and infestations) | 1 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Abdomen/GI
Insomnia (General disorders) | 7 (8) | 2 (2) | 5 (5) | 4 (5) | 7 (7) | 6 (6) | 3 (3) | 4 (4)
Involuntary Movement (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Leukocytosis (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Libido (Reproductive system and breast disorders) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypomagnesemia (Metabolism and nutrition disorders) | 1 (1) | 3 (3) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Memory Impairment (Nervous system disorders) | 9 (9) | 5 (5) | 7 (7) | 8 (9) | 8 (8) | 7 (7) | 4 (4) | 4 (4)
High Lactate Dehydrogenase (Blood and lymphatic system disorders) | 8 (10) | 3 (3) | 4 (5) | 5 (7) | 3 (3) | 3 (4) | 2 (2) | 3 (4)
High BUN Serum (Blood and lymphatic system disorders) | 5 (9) | 2 (2) | 8 (13) | 4 (6) | 6 (8) | 2 (2) | 2 (2) | 1 (1)
Hyperlipidemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
High Chloride Serum (Metabolism and nutrition disorders) | 3 (4) | 3 (6) | 5 (7) | 6 (9) | 2 (4) | 5 (9) | 2 (3) | 2 (2)
Hyperphosphatemia (Metabolism and nutrition disorders) | 4 (7) | 1 (1) | 2 (2) | 1 (1) | 3 (4) | 2 (2) | 4 (4) | 0 (0)
High Bicarbonate (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Low Chloride Serum (Metabolism and nutrition disorders) | 2 (2) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Low Protein Serum (Metabolism and nutrition disorders) | 2 (2) | 1 (2) | 3 (5) | 1 (1) | 1 (1) | 3 (6) | 2 (3) | 2 (2)
High Protein Serum (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Low Uric Acid (Metabolism and nutrition disorders) | 2 (3) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Anxiety (Nervous system disorders) | 3 (3) | 1 (1) | 3 (3) | 2 (2) | 3 (3) | 5 (5) | 4 (4) | 0 (0)
Agitation (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 2 (2) | 1 (1) | 0 (0)
Paranasal Sinus Reactions (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 11 (14) | 6 (7) | 9 (11) | 10 (12) | 11 (12) | 10 (13) | 11 (12) | 8 (8)
Neuropathy (Nervous system disorders) | 2 (2) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 1 (2) | 1 (1) — Cranial
Neuropathy - Motor (Nervous system disorders) | 1 (1) | 2 (2) | 2 (2) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Neuropathy - Sensory (Nervous system disorders) | 4 (4) | 3 (4) | 2 (2) | 2 (4) | 2 (2) | 4 (4) | 4 (4) | 4 (4)
Tingling (Nervous system disorders) | 3 (3) | 2 (2) | 0 (0) | 0 (0) | 3 (3) | 3 (3) | 4 (5) | 1 (1)
Dysesthesias (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Numbness (Nervous system disorders) | 4 (4) | 2 (2) | 3 (3) | 3 (4) | 2 (2) | 4 (5) | 7 (8) | 1 (1)
Unsteady Gait (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Radiculopathy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anopsia (Eye disorders) | 2 (2) | 2 (2) | 3 (3) | 2 (2) | 3 (3) | 4 (4) | 3 (4) | 6 (6)
Lowered Visual Acuity (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 1 (1) | 0 (0)
Loss of Vision (Eye disorders) | 2 (2) | 0 (0) | 2 (2) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Otitis (Ear and labyrinth disorders) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 2 (3) | 1 (1) | 1 (1) | 0 (0)
Chest Pain (Respiratory, thoracic and mediastinal disorders) | 5 (6) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 3 (3) | 1 (1) | 1 (1)
Ear Pain (Ear and labyrinth disorders) | 4 (5) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 2 (2) | 1 (1) | 0 (0)
Breast Pain (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Back Pain (Musculoskeletal and connective tissue disorders) | 5 (5) | 2 (2) | 1 (1) | 3 (3) | 1 (1) | 1 (1) | 1 (1) | 2 (2)
Joint Pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 2 (2) | 5 (6) | 0 (0) | 3 (4) | 0 (0) | 2 (2)
Abdomen/GI Pain (Gastrointestinal disorders) | 2 (2) | 1 (1) | 2 (2) | 5 (6) | 2 (2) | 1 (1) | 2 (2) | 4 (5)
Knee Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ankle Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Shoulder Pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 0 (0)
Jaw Pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Wrist Pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neuralgia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Suprapubic
Photophobia (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Edema (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 1 (1) — Eye
Retinopathy (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chills (General disorders) | 1 (1) | 1 (1) | 1 (1) | 2 (4) | 0 (0) | 3 (3) | 3 (3) | 0 (0)
Seizure (Nervous system disorders) | 5 (5) | 6 (6) | 5 (14) | 7 (10) | 11 (13) | 8 (12) | 8 (8) | 2 (2)
Hypernatremia (Metabolism and nutrition disorders) | 2 (3) | 2 (2) | 2 (2) | 2 (2) | 1 (1) | 3 (4) | 0 (0) | 2 (2)
Somnolence (Nervous system disorders) | 2 (2) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 3 (4) | 5 (5) | 4 (4)
Tremor (Nervous system disorders) | 2 (2) | 3 (3) | 2 (2) | 2 (2) | 2 (2) | 3 (3) | 3 (3) | 7 (7)
Tinnitus (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0) | 3 (3) | 2 (2) | 2 (2) | 1 (1) | 1 (1)
Taste Alteration (Gastrointestinal disorders) | 2 (2) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Urinary Frequency (Renal and urinary disorders) | 4 (5) | 2 (3) | 1 (1) | 5 (6) | 2 (2) | 3 (4) | 3 (3) | 2 (2)
Vital Capacity (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thrombophlebitis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Voice Changes (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 5 (5) | 4 (4) | 4 (5) | 4 (5) | 1 (1) | 4 (4) | 5 (5) | 3 (3)
Watery Eye (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Weight Gain (General disorders) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Allergy (Immune system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Penicillin
Allergy (Immune system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Iodine
Dehydration (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1)
Cushingoid (Endocrine disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Diabetes (Endocrine disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Diplopia (Eye disorders) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 3 (4) | 0 (0)
Distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dry Eye (Eye disorders) | 0 (0) | 2 (2) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 2 (2) | 1 (1)
Dry Mouth (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 4 (4) | 0 (0) | 3 (3) | 1 (1)
Edema (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 3 (3) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) — Head and Neck
Eyelid Dysfunction (Eye disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Thrush (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Mucositis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Hiccoughs (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oral Candidiasis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Irregular Menses (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Low Phenytoin (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscle Cramps (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nail Changes (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nystagmus (Eye disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 1 (1)
Orgasmic dyfunction (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mouth Sores (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hip Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Renal Pain (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Proteinuria (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 1 (1) | 3 (6) | 2 (2) | 0 (0)
Psychosis (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinus Congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Membranous Glomerulonephritis (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thrombotic Thrombocytopenic Purpura (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ulcer (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vaginal Dryness (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Varicosities (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mood Changes (Nervous system disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Stress Incontinence (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Extraocular Movement (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Acne (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ascites (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Low BUN Serum (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 1 (1) | 1 (1)
Neck Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Throat Pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (3) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Periodontal Disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin Lesion (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bilateral Ankle Swelling (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Facial Hair Growth (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 1 (1)
Toe Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sore Throat (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Infection with Normal ANC (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Prostate
Exophoria (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Esotropia (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
CN VI Palsy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Palpitations (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Supraventricular Arrhythmia-Atrial Fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypothyroidism (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 1 (1)
Erythema Multiforme (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Hyperalbuminenia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 2 (2)
Low Lactate Dehydrogenase (Blood and lymphatic system disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 2 (4) | 0 (0) | 0 (0)
Short Term Memory (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Obesity (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 3 (4) | 1 (1)
Astigmatism (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Conjunctival Infection (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Eye Pain (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 1 (1)
Photosensitivity (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Deep Vein Thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Dysuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cheilosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Dysgeusia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Indigestion (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diverticulitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ear Wax (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Asymmetrical Optic Cup (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Creatine Phosphokinase (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ecchymosis Lower Extremity (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Edema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Larynx
Fracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dystonic Meige Syndrome (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intermittent Appetite Change (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urinary Incontinence (Renal and urinary disorders) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Bilateral Hands/Feet Swelling (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Left VII CN Palsy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Disorientation (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Light Headedness (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscles Twitching (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bronchitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Uticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tympanic Membrane Perforation (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bladder Spasms (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Burn (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Restlessness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Flu-Like Syndrome (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (3) | 0 (0)
GERD (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Polyp in the Cardia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gilbert's Disease (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hemorrhoids (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (3) | 1 (1)
Burning During Urination (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gout (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hyperreflexia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Breast Tenderness (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Anisocoria (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Partial Thromboplastin Time (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tachycardia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Chest Tightness (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Low Testosterone (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ulceration (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Face and Right Ear
Wound Complication (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Non-Infectious
CO2 Serum Low (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Swollen Eyes (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Cardiac Arrhythmia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Skin Sensitivity (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Flatulence (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Flushing (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hepatic Hemangioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Anal Incontinence (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sarcoidosis (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Agraphesthesia (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Apraxia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Otosclerosis (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Osteopenia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Facial Droop (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Deep Tendon Reflexes - Limb (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) — Decreased/Increased
Necrosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — Colon/Cecum/Appendix
Kidney Stones (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cervical Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Peripheral Vascular Disease (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vein Injury (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Injection Site Reaction (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Left Hemiparesis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Thyroid Problems (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Asymptomatic Thyroid Nodule (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes